CLINICAL TRIAL: NCT04580862
Title: Incidence Postoperative Pain After Single Visit Versus Two Visit Nonsurgical Endodontic Retreatment
Brief Title: Postoperative Pain Endodontic Retreatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Muftah Mohammed Ali Akrym, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: pop rct
Record Dates: First submitted 2020-05-05; First posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Endodontically Treated Teeth
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 Non-surgical endodontic retreatment in single visit (Experimental): Single visit treatments have gained more popularity. Completing the treatment in a single appointment has many advantages including reduction in treatment time and cost, lower risk of micro leakage and recontamination of root canals between appointments
  Interventions: Other: Non-surgical endodontic retreatment in single visit
- group 2 Non-surgical endodontic retreatment in Two-visit (Active Comparator): Two-visit endodontic treatment with intra-canal medication was traditionally found to be effective in decreasing the number of flare-up in all retreatment cases and in reducing postoperative pain of previously symptomatic teeth
  Interventions: Other: Non-surgical endodontic retreatment in single visit

INTERVENTIONS:
Other: Non-surgical endodontic retreatment in single visit — Full medical and dental history using a schematic dental chart, will be obtained from all patients treated during this study.
  Other Names: Non-surgical endodontic retreatment in Two-visit

SUMMARY:
To compare the incidence of post-operative pain after single-visit versus two-visit non-surgical endodontic retreatment.

DETAILED DESCRIPTION:
Post treatment failure could be treated by two options including orthograde retreatment and apical surgery . In a previous study, orthograde retreatments presented a success rate of 81 % classified as healed and 93 % as no symptoms and fully functional. In a systematic review, it has also been concluded that endodontic surgery offers more favorable initial success but orthograde retreatment yields to a better long-term outcome . Although early results of single-visit treatments are contradictory ; Completing the treatment in a single appointment reduces the treatment time and cost, decreases micro leakage risk and avoids recontamination of root canals between appointments in multiple-visit treatments . Again, reviewing the literature concerning primary treatment showed that, no significant differences were observed in healing of periapical radiolucency between teeth treated in single-visit and those treated in two-visits. Even, after using calcium hydroxide for four weeks . The presence of a positive bacterial culture at the time of filling did not influence the outcome of treatment .

Thorough online search revealed that, few studies are found concerning post- operative pain after single visit retreatment . The present study is designed to compare the effects of single-visit and two-visit root canal treatments on postoperative pain in retreatment cases. The primary outcome measure of this study is proposed to be whether single-visit root canal retreatment influenced the occurrence of postoperative pain as compared to two-visit treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinically asymptomatic.
* Previously treated teeth in need of retreatment due to leakage and/or improper filling.
* No periapical radiolucency.
* No percussion pains.
* Age 20 - 45.
* Premolar teeth.
* Male & female.

Exclusion Criteria:

* Complicating compromised patient.
* Tenderness to percussion and acute apical abscess.
* Presence of an associated sinus tract.
* Presence of swelling in adjacent soft tissue.
* Teeth with periodontal pathologies or mobility.
* Teeth representing root fracture.
* Pregnant women.
* If analgesics or antibiotics have been administrated by the patient during the past 24 hours.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and intensity of postoperative | At one week after each visit
  Evaluate incidence and intensity of postoperative pain at 6,12,24, 48hours , and one week using numerical visual scale (NRS) after each visit endodontic retreatment

SECONDARY OUTCOMES:
Number of analgesic tablets | baseline
  Number of analgesic tablets taken by the patient after endodontic retreatment

REFERENCES:
- [Background] Erdem Hepsenoglu Y, Eyuboglu TF, Ozcan M. Postoperative Pain Intensity after Single- versus Two-visit Nonsurgical Endodontic Retreatment: A Randomized Clinical Trial. J Endod. 2018 Sep;44(9):1339-1346. doi: 10.1016/j.joen.2018.05.017. Epub 2018 Jul 24. PMID 30054099